CLINICAL TRIAL: NCT02421445
Title: An Observational Study to Characterize Human Milk From Mothers Delivering Term SGA and AGA Infants.
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 12.23 NRC
Record Dates: First submitted 2015-04-01; First posted 2015-04-20 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Small for Gestational Age (SGA) Infants; Appropriate for Gestational Age (AGA) Infants
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to characterize human milk of mothers delivering term SGA and term AGA infants. This is an observational, exploratory, longitudinal (from birth to 6 months postpartum), 4 parallel groups, and multi-centric study. Total 300 subjects will be randomised in the study assuming 20% dropout, 240 subjects will be enrolled. The recruitment period for the study in India is for 6 months.

DETAILED DESCRIPTION:
This is an observational study to characterize human milk of mothers delivering term SGA and term AGA infants. This is an observational, exploratory, longitudinal (from birth to 6 months postpartum), 4 parallel groups, and multi-centric study. Total 300 subjects will be randomised in the study assuming 20% dropout, 240 subjects will be enrolled. The recruitment period for the study in India is for 6 months.

The Primary Objective of the study is to characterize and quantify maternal milk composition from mothers of adequately nourished and under nourished status delivering term Small for Gestational Age (SGA) infants, compared to adequately-nourished and undernourished mothers delivering term Appropriate for Gestational Age (AGA) infants as defined in Fenton growth chart 2013.

The secondary objective of the study is-

1. Association of maternal milk components with dietary intake and nourishment status of the mother.
2. Associations of maternal and infant clinical parameters to maternal milk nutrients.
3. To explore and analyze additional functional milk components, such as triacylglycerol, cholesterols, carotenoids, vitamins, microbiota, peptide profile, microRNA, cytokines, growth factors and hormones.

The subject will enroll in the study after signing the Informed Consent Form after delivery the infants (i.e. term AGA & term SGA) within 72 hours. Total Duration of the study for subject is 24 weeks. Sponsor will notify the end of study after 90 days of last subject last visit. Principal Investigator responsibility is to detect and document AE and SAE

ELIGIBILITY:
Inclusion Criteria:

1. All mothers who delivered term infants, either SGA or AGA
2. Mothers between 18 and 40 years of age inclusive, at the time of enrolment
3. Having decided to predominantly breast-feed their new born baby at least until 6 months of age
4. Having permanent residence at a maximum distance of 50km from the hospital/center of investigation for the duration of this study and being able to follow all the steps of this study
5. Willing to provide informed consent according to the requirements of local regulations.

Exclusion Criteria:

1. Preterm delivery (≤ 36 weeks + 6 days completed) of gestational age)
2. Currently participating or having participated in an interventional clinical trial during the last 4 weeks prior to the beginning of this study
3. Having a BMI ≥ 25.0
4. Chewing tobacco, smoking or drinking alcohol (> 1 glass per day), consuming illicit drugs during pregnancy or/and duration of the study
5. Presenting any disease or medical condition which might prevent breast-feeding or collecting the human milk samples or for which breast-feeding is contraindicated
6. Having diabetes or gestational diabetes mellitus
7. Presenting dietary problems/illnesses such as anorexia, bulimia and celiac disease
8. Subject unable to comply with study procedures or unable to come to hospital for the study visits.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy (normal BMI) and undernourished (low BMI) women volunteers
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Maternal Milk Composition Characterization and Quantification | Visit 1 (Delivery - up to 72 hr post partum)
  Milk samples collected for analyses of functional milk components, such as macronutrients (total fat, total protein, total lactose, total energy, crude proteins and total solids) and total protein analysis by BCA kit.
Maternal Milk Composition Characterization and Quantification | Visit 2 ( 6 week )
  Milk samples collected for analyses of functional milk components, such as macronutrients (total fat, total protein, total lactose, total energy, crude proteins and total solids) and total protein analysis by BCA kit.
Maternal Milk Composition Characterization and Quantification | Visit 3 (10 Week)
  Milk samples collected for analyses of functional milk components, such as macronutrients (total fat, total protein, total lactose, total energy, crude proteins and total solids) and total protein analysis by BCA kit.
Maternal Milk Composition Characterization and Quantification | Visit 4 (14 week)
  Milk samples collected for analyses of functional milk components, such as macronutrients (total fat, total protein, total lactose, total energy, crude proteins and total solids) and total protein analysis by BCA kit.
Maternal Milk Composition Characterization and Quantification | Visit 5 (24 week)
  Milk samples collected for analyses of functional milk components, such as macronutrients (total fat, total protein, total lactose, total energy, crude proteins and total solids) and total protein analysis by BCA kit.

SECONDARY OUTCOMES:
Dietary intake | 3 consecutive days the week prior visit 2 (6 Week)
  Assessed by a dietary questionnaire and correlated to infants and mothers'characteristics.
Dietary intake | 3 consecutive days prior to visit 3 (10 Week)
  Assessed by a dietary questionnaire and correlated to infants and mothers'characteristics.
Dietary intake | 3 consecutive days prior to visit 4 (14 week)
  Assessed by a dietary questionnaire and correlated to infants and mothers'characteristics.
Dietary intake | 3 consecutive days prior to visit 5 (24 week)
  Assessed by a dietary questionnaire and correlated to infants and mothers'characteristics.
Maternal milk composition analysis | 5 visits from post delivery to 24 weeks.
  Other exploratory analyses such as fatty acids, cholesterol, phospholipids, gangliosides, oligosaccharides, peptides, amino acids, minerals, triacylglycerol, carotenoids, vitamins, microbiota, peptide profile, microRNA, cytokines, growth factors and hormones.
Associations of maternal and infant clinical parameters to maternal milk nutrients | 5 visits from post delivery to 24 weeks
  Correlation of maternal milk composition to mother's diet, stage of lactation, type of delivery, sex of the infant, single/multiple birth, infant anthropometric measures (weight, length and head circumference), gestational age at birth and birth anthropometrics.

CONTACTS AND LOCATIONS:
Overall Officials: Neelam Kler, Dr, Principal Investigator — Sir Ganga Ram Hospital, Delhi; Anil Kumar Sapare, DR, Principal Investigator — Muzumdar Shaw Medical Centre, Bengalore; Sarika Prasad, Dr, Principal Investigator — Aadithya Adhikari Hospital
Locations (3):
- India (3):
  - Muzumdar Shaw Medical Centre, Delhi, Bangalore
  - Aadithya Adhikari Hospital, Mysore, Karnataka
  - Sir Ganga Ram Hospital, New Delhi